CLINICAL TRIAL: NCT00000333
Title: Evaluation of Efficacy of Benztropine for Cocaine Craving
Brief Title: Evaluation of Benztropine for Cocaine Craving - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: NIDA-3-0009-2; Y01-3-0009-2
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2002-12

CONDITIONS: Cocaine-Related Disorders
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Benztropine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: Benztropine

SUMMARY:
The purpose of this study is to compare the efficacy of benztropine (or DA reuptake inhibitor) with atropine and placebo in affecting stimulated craving to cocaine cues.

ELIGIBILITY:
Please contact site for information.

Ages: 22 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 2001-05 (Actual); Primary Completion 2003-01 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Stimulated and non-stimulated craving

CONTACTS AND LOCATIONS:
Overall Officials: Steven Deutsch, M.D., Principal Investigator — Washington D.C. Veterans Affairs Medical Center
Locations (1):
- Washington DC VA, Washington D.C., District of Columbia, United States